CLINICAL TRIAL: NCT02869178
Title: Analysis Of Strain Myocardial Associated With The Exercise Tolerance In Patients With Heart Failure Systolic
Brief Title: Strain X Cardiopulmonary Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daniella Cunha Brandao (Other)
Responsible Party: Sponsor-Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Other Study IDs: Rafael_cardio
Record Dates: First submitted 2016-08-06; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Introduction : Patients with heart failure (HF ) with systolic dysfunction of moderate to severe exhibit significant reduction in the ability to exercise compared to those with mild dysfunction , and have worse prognosis. However, some clinical markers of severity and diagnosis widely used in this population such as ejection fraction (EF) , are not always able to translate the actual degree of cardiac damage as well as their relationship with the cardiorespiratory fitness of these individuals and prognosis .

Objective: To evaluate the ability of the global longitudinal strain ( GLS ) in predicting exercise tolerance in heart failure patients with moderate and significant systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* moderate and significant systolic dysfunction (LVEF < 45%) assessed by transthoracic echocardiography recent ( last month before evaluation ) Teichholz method , or when in the presence of contractile deficit target , by the Simpson method.

Exclusion Criteria:

* deformity in the face to prevent the coupling of the mask to perform the CPET ,
* orthopedic and neurological diseases that could make it impossible to perform the tests ,
* patients with psychiatric disorders that restricted them to respond to the questionnaire ,
* HF FC IV or hospitalization in the last three months ,
* angina unstable;
* myocardial infarction or heart surgery up to three months before the survey ;
* FEV1 / FVC <70 % predicted characterizing obstructive respiratory disorder .

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adults 21-65 years diagnosed with HF of all etiologies , in functional class II and III by the New York Heart Association ( NYHA ) , sedentary , of both sexes.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Echocardiography for obtaining the "strain " | 1 day
  To strain of technical analysis will be used echocardiography analysis software ( EchoPAC , GE Medical Systems, Horten , Norway, version 10.0 ) . The images will be analyzed in the longitudinal sections ( 4 bedrooms , 3 bedrooms and 2 cameras) . The endocardium is drawn manually from the septum to the lateral mitral annulus. A region of interest will be applied automatically by the software.

SECONDARY OUTCOMES:
Cardiopulmonary Test | 1 day
  Cardiopulmonary exercise testing will be carried out by the treadmill ramp method ( Centurium 300 , Micromed , Brazil ) through ErgoPC Elite® software associated with the electrocardiogram ( Micromed , Brazil ) with 12 channels. Respiratory variables will be evaluated by a gas analyzer ( Cortex - Metalyzer II , Germany) being obtained in standard conditions of temperature , pressure and humidity ( STPD ) , breath - by - breath , with the patient breathing in a face mask without leaks during exercise. Will be assessed during the test , functional capacity , measured in METs , VO2 , VE / VCO 2 , VE / VCO 2 slope , T1 / 2VO2 and RFC1 .

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernmabuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Becker M, Hoffmann R, Kuhl HP, Grawe H, Katoh M, Kramann R, Bucker A, Hanrath P, Heussen N. Analysis of myocardial deformation based on ultrasonic pixel tracking to determine transmurality in chronic myocardial infarction. Eur Heart J. 2006 Nov;27(21):2560-6. doi: 10.1093/eurheartj/ehl288. Epub 2006 Oct 11. PMID 17035253
- [Result] Belohlavek M, Pislaru C, Bae RY, Greenleaf JF, Seward JB. Real-time strain rate echocardiographic imaging: temporal and spatial analysis of postsystolic compression in acutely ischemic myocardium. J Am Soc Echocardiogr. 2001 May;14(5):360-9. doi: 10.1067/mje.2001.110786. PMID 11337681
- [Result] Chan J, Hanekom L, Wong C, Leano R, Cho GY, Marwick TH. Differentiation of subendocardial and transmural infarction using two-dimensional strain rate imaging to assess short-axis and long-axis myocardial function. J Am Coll Cardiol. 2006 Nov 21;48(10):2026-33. doi: 10.1016/j.jacc.2006.07.050. Epub 2006 Oct 31. PMID 17112992